CLINICAL TRIAL: NCT07130617
Title: A Phase Ib, Multicenter, Randomized, Double-blind, Placebo-controlled Parallel Group Clinical Study Evaluating the Efficacy and Safety of Megestrol Acetate Oral Suspension in Preventing Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy
Brief Title: Evaluation of the Efficacy and Safety of Megestrol Acetate in Preventing Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci158-101
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Efficacy; Safety; Megestrol Acetate; Adult Subject
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose of Megestrol Acetate Oral Suspension (Experimental)
  Interventions: Drug: Low dose of Megestrol Acetate Oral Suspension combined with standard therapy
- Medium dose of Megestrol Acetate Oral Suspension (Experimental)
  Interventions: Drug: Medium dose of Megestrol Acetate Oral Suspension combined with standard therapy
- High dose of Megestrol Acetate Oral Suspension (Experimental)
  Interventions: Drug: High dose of Megestrol Acetate Oral Suspension combined with standard therapy
- Megestrol Acetate Oral Suspension Placebo (Active Comparator)
  Interventions: Drug: Megestrol Acetate Oral Suspension Placebo combined with standard therapy

INTERVENTIONS:
Drug: Low dose of Megestrol Acetate Oral Suspension combined with standard therapy — A single dose of 312.5 mg/day, administered once daily (QD) for 7 consecutive days.
  Arms: Low dose of Megestrol Acetate Oral Suspension
Drug: Medium dose of Megestrol Acetate Oral Suspension combined with standard therapy — A single dose of 625 mg/day, administered once daily (QD) for 7 consecutive days.
  Arms: Medium dose of Megestrol Acetate Oral Suspension
Drug: High dose of Megestrol Acetate Oral Suspension combined with standard therapy — A single dose of 937.5 mg/day, administered once daily (QD) for 7 consecutive days.
  Arms: High dose of Megestrol Acetate Oral Suspension
Drug: Megestrol Acetate Oral Suspension Placebo combined with standard therapy — A single dose of 5 mL/day, administered once daily (QD) for 7 consecutive days.
  Arms: Megestrol Acetate Oral Suspension Placebo

SUMMARY:
To evaluate the efficacy of Megestrol Acetate Oral Suspension in Preventing Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy in Malignant Solid Tumor Patients

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled parallel-group study evaluates the efficacy, safety, and pharmacokinetic profile of megestrol acetate oral suspension in preventing nausea and vomiting induced by highly emetogenic chemotherapy. The trial plans to enroll 132 chemotherapy-naive malignant solid tumor patients scheduled to undergo initial single-day highly emetogenic chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of sex
2. Histologically or cytologically confirmed lung cancer
3. Expected survival ≥ 3 months
4. Female subjects of childbearing potential must have negative serum pregnancy test within 72 hours prior to randomization and must be non-lactating
5. Capable of comprehending and willingly providing signed informed consent form (ICF), and adhering to study requirements/restrictions Exclusion Criteria

1. Received or scheduled to receive concurrent radiotherapy within 7 days prior to enrollment through Day 1-8 of treatment 2. Systemic corticosteroid therapy or sedating antihistamines within 7 days prior to enrollment 3. Poorly controlled serous cavity effusions (pleural/peritoneal/pericardial) 4. Severe cardiovascular diseases within 3 months prior to enrollment 5. Participation in other clinical trials within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects Experiencing No Nausea During 0-168 Hours After Initiation of the First Chemotherapy Cycle | From 0 to 168 Hours After Initiation of Chemotherapy
Proportion of Subjects Experiencing No Nausea During 0-120 Hours After Initiation of the First Chemotherapy Cycle | From 0 to 120 Hours After Initiation of Chemotherapy

SECONDARY OUTCOMES:
Proportion of Subjects Achieving Complete Response (No significant nausea, No vomiting, etc. ) in the Acute, Delayed, Extended Delayed, 0-120 h, and 0-168 h Phases During the First Chemotherapy Cycle | From 0 to 168 Hours After Initiation of Chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PHD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China